CLINICAL TRIAL: NCT03799107
Title: The Developmental Epidemiological Study of Children Born Through Reproductive Technology
Brief Title: Developmental Epidemiological Study of Children Born Through Reproductive Technology
Acronym: DESCRT
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB 16-20474; 1R01HD084380 (NIH)
Record Dates: First submitted 2018-11-15; First posted 2019-01-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Infertility; Infertility, Female; Infertility, Male; Infertility Primary; Infertility Secondary; Infertility Unexplained
MeSH Terms: conditions — Infertility; Infertility, Female; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Children born with assistance
- Prospective: People who have sought evaluation/treatment for infertility

SUMMARY:
DESCRT will be a long-term study that both looks back in time, at successful pregnancies, and forward in time at early pregnancy and long-term as these children grow. Currently, there are limited data on the long-term effects of infertility and infertility treatments on children. There are some studies to suggest that these children may have altered metabolic profiles, but this study aims to be the largest study to answer this question.

DETAILED DESCRIPTION:
Over the past 30 years, much of the research and clinical effort in the field of ART had to do with improving outcome in terms of successful pregnancy. However, as these rates have increased, attention is slowly turning to focus on the health of the resultant child. Short-term health complications, in particular birth defects,have been well-described. However, even this "hard" outcome has been difficult to characterize as studies used different methodologies, varied age of detection, and frequently didn't have an appropriate comparison group. When underlying parental factors and infertility are included in the analyses, the association is substantially weakened or disappears completely. This exemplifies the problems with much of the currently available research regarding childhood outcomes following ART. While the health of children born through these technologies is of critical public health interest, and of personal interest to families, only limited data exist.

In order to evaluate the potential risk to long-term health of children conceived through assisted reproductive technologies (ART) and non-IVF fertility treatments (NIFT), rigorous epidemiological methods, appropriate characterization of the exposure, standardized collection of outcome data, and appropriate comparison groups are required. The proposed Developmental Epidemiological Study of Children born through Reproductive Technology (DESCRT) is aimed to carefully address these important characteristics.

ELIGIBILITY:
Retrospective arm

Inclusion criteria:

- children conceived by parent(s) who sought evaluation/treatment for infertility

Exclusion criteria:

- Children with chronic medical illnesses that prevent a study visit

Prospective arm

Inclusion criteria:

- seeking evaluation/treatment for infertility

Exclusion criteria:

- none

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective:
  - children conceived by parent(s) who sought evaluation/treatment for infertility
  Prospective:
  - people seeking evaluation/treatment for infertility
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Estimated)
Dates: Start 2017-07-14 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic testing of child - fasting glucose | 1 day at study visit
  Fasting glucose mg/dL
Metabolic testing of child - fasting insulin | 1 day at study visit
  Fasting insulin uIU/mL
Metabolic testing of child - uric acid | 1 day at study visit
  uric acid mg/dL
Metabolic testing of child - total cholesterol | 1 day at study visit
  Cholesterol, Total mg/dL
Metabolic testing of child - HDL cholesterol | 1 day at study visit
  HDL cholesterol mg/dL
Metabolic testing of child - LDL cholesterol | 1 day at study visit
  LDL cholesterol mg/dL
Metabolic testing of child - Triglycerides | 1 day at study visit
  Triglycerides mg/dL
Metabolic testing of child - cholesterol ratio | 1 day at study visit
  CHOL/HDLC ratio
Metabolic testing of child - non-HDL cholesterol | 1 day at study visit
  Non-HDL cholesterol mg/dL
Metabolic testing of child - Alanine Aminotransferase | 1 day at study visit
  Alanine Aminotransferase (ALT) U/L

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle Cedars, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adeleye AJ, Zablotska L, Rinaudo P, Huang D, Lustig RH, Cedars MI. Study protocol for a Developmental Epidemiological Study of Children born through Reproductive Technologies (DESCRT). Hum Reprod Open. 2023 May 5;2023(2):hoad013. doi: 10.1093/hropen/hoad013. eCollection 2023. PMID 37265937